CLINICAL TRIAL: NCT00610181
Title: Magnetic Resonance Imaging (MRI) for Preoperative Staging of Patients With Invasive Lobular Carcinoma of the Breast
Brief Title: Magnetic Resonance Imaging in Patients With Breast Cancer
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2007-0736
Record Dates: First submitted 2008-01-24; First posted 2008-02-07 (Estimated); Last update posted 2015-07-01 (Estimated); Status verified 2015-06

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Breast Carcinoma; Invasive Lobular Cancer; Mixed Invasive Ductal-lobular Carcinoma; Magnetic Resonance Imaging; MRI
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Breast MRI: Magnetic resonance imaging (MRI) of breast for patients with invasive lobular carcinoma of the breast.
  Interventions: Procedure: MRI

INTERVENTIONS:
Procedure: MRI — MRI of both breasts, results used for surgery, then MRI repeated in 1 year as part of routine follow-up after surgery.

SUMMARY:
The goal of this clinical research study is to learn how often magnetic resonance imaging (MRI) of the breast locates additional areas of cancer in the breast of patients with lobular cancer as well as in the breasts of young breast cancer patients (less than age 40 years). Researchers also hope to learn how often the results of the MRI changes the type of surgical treatment that is recommended and understand the costs associated with using MRI in the diagnostic process. Researchers also want to use a different way of looking at the MRI scans to learn if they can more easily learn the difference between a cyst and a tumor.

DETAILED DESCRIPTION:
At MD Anderson, patients with breast cancer routinely have mammograms and ultrasounds to measure the size and extent of cancer.

MRI of the breast is a technology that is better than mammograms and ultrasounds at locating cancer. Although MRI may locate more areas of cancer, it can sometimes falsely identify normal areas of the breast as cancerous.

Unlike ductal cancer of the breast (the most common type of breast cancer), lobular cancer is more difficult to see on mammograms and ultrasounds. Therefore, patients with lobular cancer of the breast may be best suited for MRI of the breast in order to more accurately determine the extent of the cancer. In addition, in young women, because the breast tissue is very dense, all types of breast tumors are harder to detect with mammogram and ultrasound and may be better seen with MRI.

A correct measurement of the size and extent of the cancer is important because this affects the recommendation for the type of surgery a patient may have.

Study Procedures:

If you agree to take part in this study, you will have an MRI of both breasts.

For the MRI, part or all of the body will be passed into a long, narrow tube scanner, which is open at both ends.

The MRI images will be compared with the images from your standard of care mammogram and ultrasound images. If the MRI shows abnormalities not seen on the mammogram or ultrasound and your doctor thinks it is necessary, you may have additional testing and/or a tumor biopsy. This is part of your standard of care.

The results of this additional MRI testing will be used by your surgeon to guide his/her recommendations for your surgery.

Information like your age, diagnosis, and results of your testing will be collected as part of the data analysis for this study.

No identifying information will be sent outside of MD Anderson. Your information will be stored on a password-protected computer. Information may be kept for up to 5 years after the study ends.

This is an investigational study. The investigational part of this study is the comparison of the outcome of MRI images to mammogram and ultrasound images in determining appropriate surgical therapy.

Up to 170 patients will be take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with pure invasive lobular carcinoma or mixed invasive ductal-lobular carcinoma with the ductal component not greater that 25% OR patients under the age of 40 at diagnosis, irrespective of tumor histology
2. For women with invasive lobular carcinoma, if the pathology report from the diagnostic biopsy states that they have "predominantly" lobular histology or lobular cancer with "focal" areas/nests of ductal carcinoma, these cases will automatically be assumed to have at least 75% lobular component.
3. Women with multifocal or multicentric breast cancer are eligible if any one of the biopsy confirmed tumors meets the histologic designations outlined in Inclusion criteria #1 and #2 above.
4. Must be able to complete the MR examination within 30 days of mammography and ultrasound of the breast.
5. Age >18 years
6. Surgery planned at MDACC
7. Eastern Cooperative Oncology Group (ECOG) status 0-2
8. Creatinine and glomerular filtration rate measured or calculated within 2 weeks of MRI date

Exclusion Criteria:

1. Patients receiving neoadjuvant chemotherapy
2. Patients with pacemakers
3. Patients with severe claustrophobia
4. Obese patients exceeding the equipment weight limits and/or the circumference of the MRI portal
5. Interval between MRI and conventional locoregional staging studies (mammography/breast US) greater than 30 days.
6. Known allergy to gadolinium
7. Patients with clips/prostheses/implanted devices that are not MRI compatible
8. Compromised renal function, with a measured or calculated glomerular filtration rate of less than 60 ml/min/1.73m^2.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with invasive lobular cancer of the breast.
Sampling Method: Non-Probability Sample
Enrollment: 96 (Actual)
Dates: Start 2008-01; Primary Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Change in surgical management of patients with invasive lobular carcinoma of the breast and young breast cancer patients as a result of preoperative breast MRI | 3 years (# of times MRI changes type of surgical treatment recommended)

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Bedrosian, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: The University of Texas M.D.Anderson Cancer Center — http://www.mdanderson.org